CLINICAL TRIAL: NCT07264517
Title: A Phase 2, Double-masked, Randomized, Vehicle-controlled Study Evaluating the Safety, Tolerability, and Efficacy of GRF312 5% in Participants With Dry Eye Disease
Brief Title: Evaluating the Safety, Tolerability, and Efficacy of GRF312 5% in Participants With Dry Eye Disease (DED).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC2302
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye Disease
Keywords: Phase 2; artificial tear product; primary or secondary Sjogren's syndrome; autoimmune diseases; moderate to severe dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: GRF312 5% administered b.i.d. (morning/evening) (Experimental)
  Interventions: Drug: GRF312 5%
- Group B: Vehicle administered b.i.d. (morning/evening) (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: GRF312 5% — Immune Globulin (Human), (GRF312 5% Ophthalmic Solution
  Arms: Group A: GRF312 5% administered b.i.d. (morning/evening)
Other: Placebo Comparator — Vehicle.
  Arms: Group B: Vehicle administered b.i.d. (morning/evening)

SUMMARY:
This is a Phase 2, multi-site, double-masked, randomized, vehicle-controlled, study designed to evaluate the safety, tolerability, and efficacy in adult participants with DED.

ELIGIBILITY:
Inclusion criteria 3. Participant willing and able to self-administer eye drops, follow instructions during the Run-in Period and Treatment Period, and be present for the required visits for the duration of the study.

4. Participant-reported history of DED in O.U. 5. History of non-prescription (over-the-counter) artificial tear product use within 30 days prior to start of the Screening.

7. Participants with primary or secondary Sjogren's syndrome (e.g., rheumatoid arthritis, systemic lupus erythematosuis,) or other autoimmune diseases (e.g., multiple sclerosis, inflammatory bowel disease) are eligible for enrollment consideration provided the participant meets all other inclusion and exclusion criteria, AND, is not in a medical state in the opinion of the Investigator that could interfere with study parameters, is not taking systemic/ocular steroids, and is not receiving systemic drugs to actively manage their baseline medical state.

8. Have a Current-corrected Visual Acuity (CCVA), using corrective lenses (spectacles) if necessary, in O.U. of + 0.7 or better as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) chart.

A participant must meet all the following inclusion criteria at both Screening and Randomization (Day 1) in the same eye to be eligible for participation in this study:

9. Have moderate to severe DED in at least one eye, as defined by meeting ALL the following criteria in the same eye:

* Unanesthetized STT score of > 1 and ≤ 7 mm over five minutes.
* Total corneal fluorescein staining score of ≥ 4 [0 to 15 National Eye Institute scale] 10. Have symptom severity score of ≥ 60 for Eye Discomfort on the Individual Symptom Severity Assessment VAS (0 to 100) at Screening and a Symptom Severity Score of ≥ 50 for Eye Discomfort on the Individual Symptom Severity Assessment VAS (0 to 100) at Randomization (Day 1).

Exclusion Criteria

1. Has a known hypersensitivity or contraindication to the study drug(s) or their components.
2. In the opinion of the Investigator, be unwilling or unable to comply with the study protocol or unable to successfully self-administer eye drops.
3. Use of any IP or device within 30 days prior to start of the Screening or during the study period.
4. Any ocular condition that, in the opinion of the Investigator, could affect study parameters including, but not limited to, eyelid margin disorders (e.g., significant blepharitis including staphylococcal, demodex or seborrheic; severe meibomian gland disease, excessive lid laxity, floppy eyelid syndrome, ectropion or entropion), advanced conjuctivochalasis, Salzmann's nodular degeneration, iritis, uveitis, and/or active ocular infection.
5. Participants with DED secondary to scarring (such as that seen with irradiation, alkali burns, Steven-Johnson syndrome, cicatricial pemphigoid) or destruction of conjunctival goblet cells (as with Vitamin A deficiency) are not eligible for the study. Participants with incidental scars secondary to refractive surgery (i.e., LASIK surgery) that, in the opinion of the Investigator, will not interfere with study compliance and/or outcome measures are not excluded from the study.
6. Known history of alcohol and/or drug abuse within the past 12 months, that in the opinion of the Investigator, may interfere with study compliance, outcome measures including safety parameters, and/or general medical condition of the participant.
7. History of active herpes simplex or zoster keratitis in either eye.
8. History of neurotrophic keratitis or suspected history of neurotrophic keratitis in the clinical judgement of the Investigator (e.g., abnormal Cochet-Bonnet test).
9. Intraocular pressure (IOP) > 22 mmHg at the Screening Visit.
10. Use of below listed medications and/or procedures within the appropriate pre-study period and throughout the study:

    a. Prohibited during the Screening Visit and throughout the study: i. Artificial tear substitutes ii. Current use of eye drops for glaucoma b. Prohibited 7 days prior to the Screening Visit and throughout the study: i. Contact Lenses c. Prohibited 14 days prior to the Screening Visit and throughout the study: i. Topical ocular or systemic antibiotics ii. Serum tears iii. Topical ocular non-steroidal anti-inflammatory drugs (NSAIDS) iv. Topical ocular or oral antihistamines or mast cell stabilizers v. Topical ocular or nasal vasoconstrictors. Phenylephrine to dilate is allowed.

    d. Prohibited 30 days prior to the Screening Visit and throughout the study: i. Ocular, inhaled or intranasal or dermatologic corticosteroids. This includes corticosteroids creams used anywhere on the body.

    ii. Lifitegrast iii. Perfluorohexyloctane ophthalmic solution iv. Oxymetazoline ophthalmic solution v. 0.25% lotilaner ophthalmic solution vi. Intranasal tear neurostimulation vii. Punctal cautery and short-term dissolvable punctal plugs. Permanent punctal plugs should not be in place at least 30 days prior to the Screening Visit.

    viii. Any topical ophthalmic medications (or makeup) used for eyelash growth e. Prohibited 6 weeks prior to the Screening Visit and throughout the study: i. Topical ocular cyclosporine f. Prohibited 3 months prior to the Screening Visit and throughout the study: i. Yttrium aluminum garnet-laser posterior capsulotomy or any laser ocular surgery ii. Punctal plugs that are long-term dissolvable g. Prohibited 6 months prior to the Screening Visit and throughout the study: i. Mechanical treatments for Meibomian Gland Dysfunction (MGD) including but not limited to thermal pulsation (Lipiflow or iLux), debridement of lid margin (BlephEx), thermal application (MeiBoFlo, Tear Care), or meibomian gland probing ii. Eyelid surgery iii. Ocular placement of amniotic membrane in either eye h. Prohibited 12 months prior to the Screening Visit and throughout the study: i. Any incisional intraocular surgical procedure ii. Have had incisional ocular surface surgery, including but not limited to LASIK or similar type of corneal refractive surgery and pterygium removal i. Prior history i. Use of isotretinoin ii. Corneal transplant or partial corneal transplant
11. Any significant chronic illness that, in the opinion of the Investigator, could interfere with the study parameters, including, but not limited to, severe cardiopulmonary disease, poorly controlled hypertension, and/or poorly controlled diabetes.
12. Has known previous or current infection of Hepatitis B virus (HBV), Hepatitis C virus (HCV), or Human Immunodeficiency Virus (HIV).

A participant must NOT meet the following exclusion criterion at the Randomization (Day 1) to be eligible for participation in this study:

14. Non-compliance (< 80% or > 120%) with vehicle regimen in the Run-in Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of participants with treatment-emergent AEs (TEAEs), serious TEAEs, and TEAEs leading to discontinuation. | Up to Day 84

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - GC2302 Study Site 105, Morrow, Georgia
  - GC2302 Study Site 106, Carmel, Indiana
  - GC2302 Study Site 104, Asheville, North Carolina
  - GC2302 Study Site 101, Garner, North Carolina
  - GC2302 Study Site 107, Cranberry Township, Pennsylvania
  - GC2302 Study Site 102, Memphis, Tennessee
  - GC2302 Study Site 111, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided